CLINICAL TRIAL: NCT03183401
Title: National Breast and Thyroid Screening After a Treatment Received Against a Cancer During Childhood
Acronym: DENACAPST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C 16-03
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Early Detection of Cancer
Keywords: childhood cancer survivor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DENACAPST programme represents an important initiative to provide near nation-wide roll-out of an important cancer surveillance program for childhood cancer survivors. The program is based on internationally recognized standards in cancer surveillance, which were developed by the International Guideline Harmonization Group (IGHG) with support of all relevant stakeholders in cancer survivorship research and clinical work in Europe, Canada and the United States and recognized French recommendations about breast screening for women at high risk of cancer.

With this programme, French centers organized themselves to provide to childhood cancer survivors adequate medical attention, which includes close medical surveillance for breast/thyroid cancer where appropriate, based on adequate risk stratification.

The aim of the study is to analyze if the recommendations about breast and thyroid cancer screening are followed in this population and secondly to provide more informations about these second cancers and about the screening.

DETAILED DESCRIPTION:
Every center which has patient at risk can participate. Main inclusion criteria : French childhood cancer survivor (5 years or more of delay with the treatment) - becoming adult - with a past history of radiotherapy at the age of 20 years or before, with a significant dose irradiation on the thyroid or the breast

The inclusion of patients are validated by one team

Thyroid screening programme is based on US each 2 years Breast screening programme is based mainly on MRI each year

ELIGIBILITY:
Inclusion Criteria:

* childhood cancer survivor, and
* treated with radiotherapy
* health status compatible, and
* have had a long-term follow-up consultation describing a personalized post-cancer plan and,
* informed consent signed by patient

  + Inclusion criteria for breast screening
* being a woman and being 25 years or more for breast cancer screening, with a minimum delay of 8 years after radiotherapy, or
* with a significant irradiation dose to the breast (Irradiation that delivered at least 10 Gy on at least part of the breast (v 5> 10 Gy) or on the mammary bud (v 100> 10 Gy) - (centrally validated dose) or received TBI (Total Body Irradiation)> 8 Gy according to a bi-fractioned scheme or> 6 Gy in single dose)

  +Inclusion criteria for thyroid screening:
* being a man or a woman and being 18 years or more for thyroid cancer screening with a minimum delay of 5 years after radiotherapy, and,
* with a significant irradiation dose to the thyroid (Irradiation having delivered at least 3 Gy on the thyroid (v100> 3 Gy), or having received a TBI (Total Body Irradiation)> 2 Gy, and / or treatment with 131i-metaiodobenzylguanidine), and

Exclusion Criteria:

* life expectancy <10 years due to other pathology
* patient in regular follow-up within the framework of a genetic susceptibility (ex li fraumeni)
* person placed under safeguard of justice

  + exclusion criteria for breast cancer screening :
* patient treated with bilateral mastectomy, or
* patient being treated for breast cancer, or
* patient initially treated with radiotherapy for breast cancer

  + exclusion criteria for breast cancer screening :
* Thyroidectomy, or
* patient undergoing treatment or with a personal history of thyroid cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients from FCCSS cohort / LEA cohort - or not involved in a cohort living in France treated for a malignant illness (cancer, leukemia) at the age of 20 or before ans still alive 5 years after
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-07-09 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
follow of cancer screening recommendations | 2 years
  number of persons at risk found percentage of persons at risk contacted who answered percentage of persons contacted, who answered, who accepted the screening

SECONDARY OUTCOMES:
description of thyroid cancer screening | 2 years
  evaluation of the programme
description of breast cancer screening | 2 years
  evaluation of the programme
description of second cancers | 2 years
  analyze of the histological data
psycho social analyze | 2 years
  evaluated by auto-questionaries :initial / final and comparison with persons who accepted to answer but who did not accept the screening

CONTACTS AND LOCATIONS:
Overall Officials: charlotte demoor-goldschmidt, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; florent de vathaire, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; gerard michel, Study Chair — chu; pascal auquier, Study Chair — medical university of Marseille
Locations (1):
- Charlotte Demoor-Goldschmidt, Villejuif, France

IPD SHARING:
Plan to Share IPD: No